CLINICAL TRIAL: NCT05735808
Title: A Pilot Study of the Feasibility and Non-inferiority of Patient Education About Arterial Hypertension in Virtual Reality
Brief Title: VR Education in Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poliklinika Agel, Dopravni zdravotnictvi a.s. (Other)
Responsible Party: Principal Investigator, Bogna Jiravska Godula, PI, Poliklinika Agel, Dopravni zdravotnictvi a.s.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAgel
Record Dates: First submitted 2023-01-12; First posted 2023-02-21 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Arterial Hypertension
Keywords: virtual reality education
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart physicain based education (Active Comparator): In this arm, patient education will be conducted by the physician as the gold standard.
  Interventions: Behavioral: Physician based education
- VR based education (Experimental): In this arm, patient education will be performed using 3D educational material presented in VR glasses.
  Interventions: Behavioral: VR based education

INTERVENTIONS:
Behavioral: Physician based education — Regular education provided by physician
  Arms: Standart physicain based education
Behavioral: VR based education — VR based education
  Arms: VR based education

SUMMARY:
The aim of this study is to compare standard education with VR augmented education in patients with arterial hypertension

DETAILED DESCRIPTION:
To demonstrate the technical and organizational feasibility of patient education about arterial hypertension in virtual reality. Demonstrate the non-inferiority of education conducted in virtual reality to traditional face-to-face education by a physician. To define the cost-effectiveness of education in virtual reality in the reality of progressing shortage of human resources.

Patients diagnosed with arterial hypertension as part of a routine examination in an internal medicine outpatient clinic will be randomized to education about the disease directly by a physician in one arm or using a 3D movie in VR glasses filmed by a physician in an identical outpatient clinic setting. It will be concluded by questionnaire method to compare the outcome of both education namely subjective satisfaction and objectively by using questions to evaluate the success of the education.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients with arterial hypertension

Exclusion Criteria:

* visual impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Non-Inferiority of VR augmented education: physician assessment of objective patient understanding | 18 months
  After the education, the patient will answer a prepared list of questions on arterial hypertension whose answers were mentioned in the previous education and the percentage of correct/wrong answers will be compared in both arms of the study.
Non-Inferiority of VR augmented education:subjective evaluation of education by the patient | 18 months
  After the education, the patient will rate how he/she subjectively perceived the subjective pleasantness of the education on a scale of 1 to 5 ( 1 best/ 5 worst).

CONTACTS AND LOCATIONS:
Overall Officials: Otakar Jiravsky, Study Chair — Nemocnice AGEL Trinec-Podlesi a.s.
Locations (1):
- Poliklinika Agel, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No
Only basic demographic data will be shared